CLINICAL TRIAL: NCT02526407
Title: The Impact of Creative Interventions on Symptoms of Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Music (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SATB2015
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Depression, Postpartum
Keywords: postnatal depression; mental wellbeing; baby blues; mothers; music; alternative therapies
MeSH Terms: conditions — Depression, Postpartum | interventions — Singing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Participants continue with usual care. No planned intervention.
- Group play (Active Comparator): Participants take part in 10 weeks of group play activities for one hour per week with their baby in a community setting alongside any usual care they may be receiving.
  Interventions: Behavioral: Group play
- Singing (Experimental): Participants take part in 10 weeks of group singing activities for one hour per week with their baby in a community setting alongside any usual care they may be receiving.
  Interventions: Behavioral: Singing

INTERVENTIONS:
Behavioral: Singing — Sessions will be led by a professional practitioner assisted by students from the Royal College of Music. Participants will learn songs with their babies and help to create new musical material together.
  Arms: Singing
Behavioral: Group play — Sessions will be led by a professional practitioner assisted by students from the Royal College of Music. Participants will take part in group play activities.
  Arms: Group play

SUMMARY:
Post-natal depression (PND) is anticipated to affect 12.9% of new mothers with at least 75,000 cases per year in the UK alone. However, despite this, there is currently a worrying lack of support for new mothers, with data suggesting that 64% of healthcare trusts in the UK do not have a strategy for treating postnatal depression, and flaws in the current pharmacological and psychological treatment models. Consequently, research into promising psychosocial interventions such as music is critical to developing new paradigms for treating postnatal depression.

This project is an ambitious programme of research that investigates the effects of music on postnatal depression through two phases: a questionnaire study and an intervention study. This record is for the intervention study. The questionnaire study has a separate record. We are accepting host hospital sites for both.

DETAILED DESCRIPTION:
The study tests the effectiveness of singing interventions led by the Royal College of Music at Chelsea and Westminster Hospital as a psychosocial tool to reduce the occurrence and effects of postnatal depression. It triangulates psychological, physiological, and biological data in a randomised control design to provide a comprehensive insight into the intervention's effects in comparison to a more common psychosocial intervention for new mothers (play groups) and a control group of no psychosocial interventions. The study aims to recruit 50-80 women into each of the three interventions (150-240 total).

The study will used a mixed-method methodology comprising validated psychological scales, in-depth qualitative interviews and observations and biomarker analysis. If results are promising, there are plans in place to scale the singing intervention to more hospitals and community settings.

Phase B will be open to NHS sites within the region of Chelsea and Westminster Hospital London from which women could travel to the sessions to take part.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a child up to 9 months old
* Symptoms suggestive of PND at a minimum score of 10 on the EPDS

Exclusion Criteria:

* Outside the limits of the number of weeks pregnant/post birth
* Living outside England
* Refusal to participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Postnatal depression | Change from baseline at 6 weeks and 10 weeks
  Measured with the Edinburgh Postnatal Depression Scale

SECONDARY OUTCOMES:
Mental wellbeing | Change from baseline at 6 weeks and 10 weeks
  Measured with the short Warwick-Edinburgh Mental Wellbeing Scale
Self-esteem | Change from baseline at 6 weeks and 10 weeks
  Measured with the Rosenberg Self-esteem scale
Social functioning | Change from baseline at 6 weeks and 10 weeks
  Measured with the Social Provisions Scale
Inflammatory immune response | Change from baseline at 6 weeks and 10 weeks
  Measured with saliva samples to test for cortisol and cytokine activity

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Williamon, PhD, Study Chair — Royal College of Music / Imperial College London
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital, London
  - Centre for Performance Science, Royal College of Music, London

REFERENCES:
- [Derived] Fancourt D, Perkins R. Creative interventions for symptoms of postnatal depression: A process evaluation of implementation. Arts Health. 2019 Feb;11(1):38-53. doi: 10.1080/17533015.2017.1413398. Epub 2018 Jan 23. PMID 31038038
- [Derived] Perkins R, Yorke S, Fancourt D. How group singing facilitates recovery from the symptoms of postnatal depression: a comparative qualitative study. BMC Psychol. 2018 Aug 17;6(1):41. doi: 10.1186/s40359-018-0253-0. PMID 30119704
- [Derived] Fancourt D, Perkins R. Effect of singing interventions on symptoms of postnatal depression: three-arm randomised controlled trial. Br J Psychiatry. 2018 Feb;212(2):119-121. doi: 10.1192/bjp.2017.29. PMID 29436333